CLINICAL TRIAL: NCT02096874
Title: The Effect of Bevacizumab on Peripheral Retinal Changes as Imaged by Wide -Field Fluorescein Angiography in Diabetic Macular Edema
Brief Title: Bevacizumab and Peripheral Retinal Changes on Wide Field Angiography in Diabetic Macular Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Khaled Eye Specialist Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP 1310
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Non-proliferative Diabetic Retinopathy; Proliferative Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Peripheral retinal ischemia; ultra wide field fluorescein angiography; Bevacizumab
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Other): Each study subject will recieve Intravitreal injection of 1.25mg/0.05 cc each 5 weeks for the first 3 months then PRN for six month.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Intravitreal injection of 1.25mg/0.05 cc each 5 weeks for the first 3 months then PRN for six month
  Other Names: Avastin

SUMMARY:
Ultra-wide field fluorescein angiography can detect the response of anti VGEF therapy such as Avastin on retinal ischemia in the setting of diabetic macular edema.

DETAILED DESCRIPTION:
The major causes of vision loss in diabetic retinopathy are diabetic macular edema (DME) characterized by thickening of the macula due to abnormal leakage of the retinal vasculature. Ischaemic changes and microvascular pathologies have long been hypothesized to play a role in the development of DME. In diabetic retinopathy, ischaemia stimulates the production of vascular endothelial growth factor (VEGF), which can lead to the breakdown of blood-retinal barriers, and may cause DME through an increase in retinal vessel permeability. DME is best evaluated by optical coherence tomography (OCT) while retinal ischemia is determined by Fluorescein angiography. With the avaiability of ultra wide field fluorescein angiography, the investigators can now accurately measure the degree of ischemia in peripheral retina. Thus, this study will provide us data on the degree of retinal ischemia in nonproliferative diabetic retinopathy (NPDR) and proliferative diabetic retinopathy (PDR) cases as well as the measurable change that occurs in retinal ischemia after intra vitreal injection of bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic patients at age >18year with DME
2. Scheduled for Avastin therapy
3. Adequate media to obtain OCT and UWFA

Exclusion Criteria:

1. Macular pathology of any etiology
2. Preexisting systemic disease causing retinal ischemia
3. Previous laser or anti-VEGF treatment in past 3 months
4. Previous retina surgery in past 2 months
5. Allergy to fluorescein dye
6. Psychiatric disorder, Alzheimer disease and Dementia or any other disorder precluding follow-up or continuation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Peripheral retinal ischemia | 24 weeks
  Change in peripheral retinal ischemia after intravitreal bevacizumab injection in non proliferative diabetic retinopathy and proliferative diabetic retinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Saba al Rashaed, MD, Principal Investigator — King Khaled Eye Specialist Hospital
Locations (1):
- King Khaled Eye Specialist Hospital, Riyadh, Saudi Arabia